CLINICAL TRIAL: NCT04160442
Title: Use of a Patient Preferences Shared Decision-Making Encounter Tool in Clinical Practice for Patients With DLBCL and FL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carevive Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 419 NHL SDM
Record Dates: First submitted 2019-11-01; First posted 2019-11-13 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Diffuse Large B Cell Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Carevive CarePlanning System — Subject will complete brief survey prior to seeing provider in clinic. Utilizing the CarePlanning System, the provider will review the subject's responses directing the conversation and treatment decision will be made. A treatment careplan will be developed and given to the subject.

SUMMARY:
The goal of this project is to test the feasibility of a Patient Preferences in Shared Decision-Making encounter tool (PPSDM) in the clinical context of Diffuse Large B-Cell Lymphoma (DLBCL) and Follicular Lymphoma (FL). This project will evaluate the feasibility of a shared decision-making (SDM) model that employs an "encounter tool"1 to facilitate SDM at the point of a treatment decision for patients with DLBCL and FL.

DETAILED DESCRIPTION:
This project is a single-arm pilot project conducted with 90 patients with newly diagnosed or recurrent DLBCL or FL and their providers at three medical oncology practices. Utilizing the PPSDM tool in the Carevive electronic platform, patients will report their needs, preferences, values and goal prior to the treatment decision-making focused clinical encounter. The treating provider will receive the patient results prior to the visit and can use these to facilitate SDM in treatment selection during the clinical encounter. Post-encounter, patients and providers will complete measures designed to assess feasibility and utility of SDM intervention. Patients will also complete measures to assess patient satisfaction with the treatment decision, patient activation, and patient perceived achievement of desired role in shared decision making and satisfaction with care.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be 18 years of age or older.
* Patient participants must have a diagnosis of new or recurrent DLBCL or FL
* All participants must be able to understand English.

Exclusion Criteria:

* Any patient who cannot understand written or spoken English.
* Any prisoner and/or other vulnerable persons as defined by NIH (45 CFR 46, Subpart B, C and D).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-01-16 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Satisfaction of using the Carevive treatment planning system in shared decision making will be collected from both patient and provider perspectives: questionnaires | 3 months
  patient and providers will complete questionnaires at each clinic visit. These questions will determine their satisfaction with the treatment care planning system.

SECONDARY OUTCOMES:
Evaluation of patient satisfaction and perceived shared decision making utilizing surveys at each clinic visit | 3 months
  Questionnaires answering questions regarding patient satisfaction with the treatment decision, patient activation, and patient perceived achievement of desired role in shared decision making following the technology-facilitated SDM intervention and compare differences in scores between the enrolled subjects. These surveys are part of the Carevive treatment planning platform and collect the information at each clinic visit.

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Wujcik, PhD,RN, Principal Investigator — Carevive Systems, Inc.
Locations (1):
- University of Alabama Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No